CLINICAL TRIAL: NCT00006032
Title: A Phase II Study of Intensive-Dose Topotecan, Ifosfamide/Mesna and Etoposide (TIME) Followed by Autologous Stem Cell Rescue in Metastatic Breast Cancer
Brief Title: Combination Chemotherapy Followed by Peripheral Stem Cell Transplantation in Treating Women With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: MCC-12220; MCC-12220; MCC-IRB-5699; NCI-G00-1809
Record Dates: First submitted 2000-07-05; First posted 2004-04-02 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Etoposide; Ifosfamide; Topotecan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: etoposide
Drug: ifosfamide
Drug: topotecan hydrochloride
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by autologous peripheral stem cell transplantation in treating women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy and toxicity of high dose topotecan with ifosfamide and etoposide followed by autologous peripheral blood stem cell rescue in women with metastatic breast cancer. II. Evaluate the response rates, progression free survival, engraftment, and nonrelapse related mortality in women treated with this regimen. III. Evaluate the pharmacokinetic profile of high dose topotecan with respect to the efficacy and toxicity of ifosfamide and etoposide in these women.

OUTLINE: Peripheral blood stem cells (PBSC) are harvested from the patient and stored. Patients receive ifosfamide IV over 2 hours and topotecan IV over 30 minutes on days -8 to -6, and etoposide IV daily over 24 hours on days -5 to -3. Autologous PBSC are reinfused on day 0. Patients are followed at 1, 3, 6, and 12 months, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic breast cancer that has demonstrated at least partial response to any salvage regimen Partial response defined as at least 50% reduction in measurable or evaluable disease for at least 4 weeks, no disease progression, no new lesions, or bone lesions that remain static for at least 8 weeks with an improvement in pain symptoms No more than 3 organs involved with metastatic disease No prior or active CNS involvement Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 to 64 Sex: Female Menopausal status: Not specified Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT or SGPT no greater than 2.5 times upper limit of normal No history of severe hepatic dysfunction Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No severe cardiac dysfunction Ejection fraction at least 50% by MUGA No major heart disease Controlled hypertension allowed Pulmonary: DLCO at least 50% of normal OR No symptomatic obstructive or restrictive disease Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective barrier contraception No uncontrolled insulin dependent diabetes mellitus No uncompensated major thyroid or adrenal dysfunction No significant skin breakdown from tumor or other disease No other prior malignancy in past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix No active infections HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No more than 2 prior salvage regimens for metastatic disease No prior topotecan Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: No concurrent nitroglycerin preparations for angina No concurrent antiarrhythmics for major ventricular arrhythmias

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2000-03; Primary Completion 2001-04 (Actual); Study Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen K. Fields, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States